CLINICAL TRIAL: NCT00516438
Title: A Phase I, Open-Label, Study of the Safety and Tolerability of KU-0059436 and Topotecan in the Treatment of Patients With Advanced Solid Tumours
Brief Title: Study to Assess the Safety and Tolerability of a PARP Inhibitor in Combination With Topotecan
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: KuDOS Pharmaceuticals Limited (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KU36-93; D0810C00006
Record Dates: First submitted 2007-08-13; First posted 2007-08-15 (Estimated); Last update posted 2010-12-08 (Estimated); Status verified 2010-12

CONDITIONS: Malignant Solid Tumors
Keywords: malignant solid tumours; Poly(ADP ribose); polymerases
MeSH Terms: interventions — olaparib; Topotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): Topotecan + KU-0059436
  Interventions: Drug: KU-0059436 (AZD2281)(PARP inhibitor); Drug: Topotecan

INTERVENTIONS:
Drug: KU-0059436 (AZD2281)(PARP inhibitor) — oral
  Other Names: Olaparib
Drug: Topotecan — intravenous infusion
  Other Names: Hycamtin®; Topotecan hydrochloride

SUMMARY:
The purpose of this study is to identify a safe and tolerable dose of the drug KU-0059436 that can be given in combination with topotecan chemotherapy in patients with advanced solid tumours

ELIGIBILITY:
Inclusion Criteria:

* Histological or cytological diagnosis of advanced solid tumour for which no suitable effective therapy exists;
* Evaluable disease
* Adequate bone marrow, hepatic and renal function

Exclusion Criteria:

* Any chemotherapy, radiotherapy ( except palliative), endocrine or immunotherapy within 4 weeks prior to entry; major surgery with 4 weeks of entering the study
* Heavily pre treated patient > 2 previous chemotherapy regimens for metastatic disease
* Co-existing active infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2007-07; Primary Completion 2009-03 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
To establish the maximum tolerated dose (MTD) of KU 0059436 in combination with topotecan | assessed at each visit

SECONDARY OUTCOMES:
To identify the dose limiting toxicity of the combination therapy | assessed at each visit

CONTACTS AND LOCATIONS:
Overall Officials: James Cassidy, Principal Investigator — Beaston Oncology Centre, Glasgow, UK; James Carmichael, BSc MBChB MD FRCP, Study Director — KuDOS Pharmaceutical Ltd
Locations (3):
- United Kingdom (3):
  - Research Site, Glasgow
  - Research Site, Leicester
  - Research Site, Manchester